CLINICAL TRIAL: NCT03636906
Title: A Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK Biologicals' RSV Investigational Vaccine Based on Viral Proteins Encoded by Chimpanzee-derived Adenovector (ChAd155-RSV) (GSK3389245A) in Infants
Brief Title: Respiratory Syncytial Virus (RSV) Investigational Vaccine in Infants Aged 6 and 7 Months Likely to be Unexposed to RSV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 204894; 2018-000431-27 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Safety; Respiratory syncytial virus (RSV); Vaccine; Reactogenicity; Immunogenicity; Infants
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4CMenB vaccine; PHiD-CV vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RSV1D Pooled Group (Experimental): Subjects received the interventions as follows:
  * Either 1 dose of experimental RSV (GSK3389245A) lower dose formulation at Day 1, followed by 1 dose of Placebo at Day 31 and any one the following active comparators: 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Day 61 and at the end of RSV season 1) or 3 doses of GSK's multicomponent meningococcal B vaccine or Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine or GSK's pneumococcal polysaccharide conjugate vaccine (administered at Days 61, 121 and at the end of RSV season 1).
  * Or 1 dose of experimental RSV (GSK3389245A) lower dose formulation at Day 1, followed by 1 dose of Placebo at Day 31.
  Interventions: Biological: RSV (GSK3389245A) lower dose formulation vaccine; Biological: GSK's multicomponent meningococcal B vaccine; Biological: Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine; Biological: GSK's pneumococcal polysaccharide conjugate vaccine; Biological: GSK's meningococcal group A, C, W-135 and Y conjugate vaccine; Drug: Placebo
- RSV2D Pooled Group (Experimental): Subjects received the interventions as follows:
  * Either 2 doses of experimental RSV (GSK3389245A) higher dose formulation (administered at Day 1 and Day 31) and followed by any one the following active comparators: 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Day 61 and at the end of RSV season 1) or 3 doses of GSK's multicomponent meningococcal B vaccine or Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine or GSK's pneumococcal polysaccharide conjugate vaccine (administered at Days 61, 121 and at the end of RSV season 1).
  * Or 2 doses of experimental RSV (GSK3389245A) higher dose formulation administered at Day 1 and Day 31.
  Interventions: Biological: RSV (GSK3389245A) higher dose formulation vaccine; Biological: GSK's multicomponent meningococcal B vaccine; Biological: Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine; Biological: GSK's pneumococcal polysaccharide conjugate vaccine; Biological: GSK's meningococcal group A, C, W-135 and Y conjugate vaccine
- Comparator_Placebo Pooled Group (Active Comparator): Subjects received either one of interventions schedules as follows:
  * 3 doses of GSK's multicomponent meningococcal B vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
  * 3 doses of Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
  * 3 doses of GSK's pneumococcal polysaccharide conjugate vaccine (administered at Days 31, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Day 1 and Day 121).
  * 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Day 31 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 1 and 61) .
  * 2 doses of Placebo alone (administered at Days 1 and 31).
  Interventions: Biological: GSK's multicomponent meningococcal B vaccine; Biological: Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine; Biological: GSK's pneumococcal polysaccharide conjugate vaccine; Biological: GSK's meningococcal group A, C, W-135 and Y conjugate vaccine; Drug: Placebo

INTERVENTIONS:
Biological: RSV (GSK3389245A) lower dose formulation vaccine — 1 dose of RSV (GSK3389245A) lower dose formulation vaccine administered intramuscularly at Day 1.
  Arms: RSV1D Pooled Group
Biological: RSV (GSK3389245A) higher dose formulation vaccine — 2 doses of RSV (GSK3389245A) higher dose formulation vaccine administered intramuscularly, at Day 1 and Day 31.
  Arms: RSV2D Pooled Group
Biological: GSK's multicomponent meningococcal B vaccine — 3 doses of GSK's multicomponent meningococcal B vaccine administered intramuscularly, at Day 61, Day 121 and at the end of RSV season 1, or at Day 1, Day 61 and end of RSV season 1, depending on the vaccination schedule.
  Other Names: Bexsero
Biological: Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine — 3 doses of Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine administered intramuscularly, at Day 61, Day 121 and at the end of RSV season 1, or at Day 1, Day 61 and end of RSV season 1, depending on the vaccination schedule.
  Other Names: Nimenrix
Biological: GSK's pneumococcal polysaccharide conjugate vaccine — 3 doses of GSK's pneumococcal polysaccharide conjugate vaccine administered intramuscularly, at Day 61, Day 121 and at the end of RSV season 1, or at Day 31, Day 61 and end of RSV season 1, depending on the vaccination schedule.
  Other Names: Synflorix
Biological: GSK's meningococcal group A, C, W-135 and Y conjugate vaccine — 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine administered intramuscularly, at Day 61 and at the end of RSV season 1, or at Day 31 and end of RSV season 1, depending on the vaccination schedule.
  Other Names: Menveo
Drug: Placebo — 1 dose or 2 doses of Placebo administered intramuscularly at Day 31, or at Day 1 and Day 31, or at Day 1 and Day 61, or at Day 31 and Day 121, depending on the vaccination schedule.
  Arms: Comparator_Placebo Pooled Group; RSV1D Pooled Group

SUMMARY:
The purpose of this study is to provide critical information on the safety, reactogenicity and immunogenicity profile of the investigational recombinant chimpanzee adenovirus Type 155-vectored RSV (ChAd155-RSV) vaccine in infants likely to be unexposed to RSV and will assess a single lower dose and a higher two dose regimen, before moving to future studies. This study will also assess if there is a risk of 'vaccine-induced enhanced RSV disease' after vaccination of these infants with the ChAd155-RSV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* A male or female between and including 6 and 7 months of age (from the day the infant becomes 6 months of age until the day before the infant achieves 8 months of age) at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term with a minimum birth weight of 2.5 kilograms (kg).
* Subjects' parent(s)/LAR(s) need to have access to a consistent mean of telephone contact or computer.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine. For corticosteroids, this will mean prednisone ≥ 0.5 milligrams (mg)/kg/day (for pediatric subjects), or equivalent. Topical steroids are allowed.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of scheduled routine pediatric vaccines. Scheduled routine pediatric vaccines may be administered ≥ 7 days before a dose of study vaccine or ≥ 7 days following a dose of study vaccine, with the exception of live viral vaccines which may be administered ≥ 14 days before a dose or ≥ 7 days after a dose.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* A history of, or on-going confirmed RSV disease or highly compatible clinical picture.
* Serious chronic illness.
* Major congenital defects.
* History of any neurological disorders or seizures.
* History of or current autoimmune disease.
* History of recurrent wheezing in the subject's lifetime.
* History of chronic cough.
* Previous hospitalization for lower respiratory illnesses.
* Previous, current or planned administration of Synagis (palivizumab).
* Neurological complications following any prior vaccination.
* Born to a mother known or suspected to be Human Immunodeficiency Virus (HIV)-positive .
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination .
* Family history of congenital or hereditary immunodeficiency.
* Previous vaccination with a recombinant simian or human adenoviral vaccine.
* History of any reaction or hypersensitivity to any component of the vaccines (investigational or control) or placebo used in this study or any contraindication to them.
* Hypersensitivity to latex.
* Current severe eczema.
* Acute disease and/or fever at the time of enrolment (Visit 1).
* Any clinically significant Grade 1 or any ≥ Grade 2 hematological or biochemical laboratory abnormality detected at the last screening blood sampling.
* Any medical condition that in the judgment of the investigator would make intramuscular (IM) injection unsafe.
* Any other conditions that the investigator judges may interfere with study procedures, findings.
* Any conditions that could constitute a risk for the subjects while participating to this study.
* Weight below the fifth percentile of the local weight-for-age curve according to the World Health Organization (WHO) weight- for- age tables. Participating in another clinical study, at any time during the study period, in which the subject or mother (if breastfeeding) has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Planned move to a location that will prohibit participating in the trial until study end.
* For Thailand only, subjects who have received Synflorix prior to enrolment.

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (4):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
- Brazil (2):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Ribeirão Preto, São Paulo
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec
- GSK Investigational Site, Cali, Colombia
- Finland (3):
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- GSK Investigational Site, Rome, Lazio, Italy
- GSK Investigational Site, México, Mexico
- Panama (2):
  - GSK Investigational Site, Chiriquí
  - GSK Investigational Site, Panama City
- Poland (5):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (6):
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Kayseri
- United Kingdom (2):
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Saez-Llorens X, Norero X, Mussi-Pinhata MM, Luciani K, de la Cueva IS, Diez-Domingo J, Lopez-Medina E, Epalza C, Brzostek J, Szymanski H, Boucher FD, Cetin BS, De Leon T, Dinleyici EC, Gabriel MAM, Ince T, Macias-Parra M, Langley JM, Martinon-Torres F, Ramet M, Kuchar E, Pinto J, Puthanakit T, Baquero-Artigao F, Gattinara GC, Arribas JMM, Ramos Amador JT, Szenborn L, Tapiero B, Anderson EJ, Campbell JD, Faust SN, Nikic V, Zhou Y, Pu W, Friel D, Dieussaert I, Lopez AG, McPhee R, Stoszek SK, Vanhoutte N. Safety and Immunogenicity of a ChAd155-Vectored Respiratory Syncytial Virus Vaccine in Infants 6-7 Months of age: A Phase 1/2 Randomized Trial. J Infect Dis. 2024 Jan 12;229(1):95-107. doi: 10.1093/infdis/jiad271. PMID 37477875

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analysis of this study results were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating counties rather than randomization to each of the groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Period: Overall Study
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Started | 65 | 71 | 65
Completed | 61 | 71 | 60
Not Completed | 4 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — CONSENT WITHDRAWAL, NOT DUE TO AN ADVERSE EVENT AND/OR A SERIOUS ADVERSE EVENT | 2 | 0 | 1
Not completed — NOT WILLING TO PARTICIPATE THIS VISIT | 1 | 0 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis of this study results were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating counties rather than randomization to each of the groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group | Total
Number analyzed (Participants) | 65 | 71 | 65 | 201
Age, Continuous [Mean (Standard Deviation); unit: MONTHS] | 6.4 (0.5) | 6.5 (0.5) | 6.5 (0.5) | 6.5 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 31 | 96
  Male | 33 | 38 | 34 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 1 | 2 | 4
  ASIAN | 1 | 1 | 1 | 3
  BLACK OR AFRICAN AMERICAN | 0 | 1 | 0 | 1
  OTHER, Not specified | 25 | 29 | 25 | 79
  WHITE | 38 | 39 | 37 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs) During a 7-day Follow-up Period After the First Vaccination (Administered at Day 1)
Description: Assessed solicited local AEs are erythema, pain and swelling at injection site. Any = occurrence of the adverse event regardless of intensity grade. Any redness and swelling = adverse event reported with a surface diameter greater than 0 millimeters. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, active comparators pooled and placebo groups separately to compare the expected adverse events observed from routine pediatric vaccines (active comparators) with the investigational RSV vaccine. Placebo was not pooled with active comparators as no significant difference was expected in AEs when placebo was pooled with active comparators. As pre-specified in the protocol, the choice of active comparator or placebo was based on each participating country's standard of care.
Time Frame: During a 7-day follow-up period after the first vaccination (administered at Day 1)
Population: Analysis was performed on the Exposed set, which included all subjects with at least 1 study vaccine administration documented and diary card completed after first vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Group: Subjects received 2 doses of Placebo alone (administered at Days 1 and 31).
- Active Comparators Pooled Group: Subjects received either one of interventions schedule as follows:
  * 3 doses of GSK's multicomponent meningococcal B vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
  * 3 doses of Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
  * 3 doses of GSK's pneumococcal polysaccharide conjugate vaccine (administered at Days 31, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Day 1 and Day 121).
  * 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Day 31 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 1 and 61) .
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Placebo Group | Active Comparators Pooled Group
Number analyzed (Participants) | 65 | 71 | 22 | 42
Participants
  Any Erythema | 5 | 6 | 0 | 22
  Any Pain | 11 | 10 | 1 | 17
  Any Swelling | 2 | 3 | 2 | 11

2. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs) During a 7-day Follow-up Period After the Second Vaccination (Administered at Day 31)
Description: Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, active comparators pooled and placebo groups separately to compare the expected adverse events observed from routine pediatric vaccines (active comparators) with the investigational RSV vaccine. Placebo was not pooled with active comparators as no significant difference was expected in AEs when placebo was pooled with active comparators. As pre-specified in the protocol, the choice of active comparator or placebo was based on each participating country's standard of care.
Time Frame: During a 7-day follow-up period after the second vaccination (administered at Day 31)
Population: Analysis was performed on Exposed set, which included all subjects with at least 1 study vaccine administration documented and diary card completed after second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Placebo Group | Active Comparators Pooled Group
Number analyzed (Participants) | 63 | 71 | 20 | 41
Participants
  Any Erythema | 8 | 7 | 0 | 11
  Any Pain | 5 | 9 | 0 | 6
  Any Swelling | 1 | 3 | 0 | 6

3. Primary Outcome: Number of Subjects With Any Solicited General AEs During a 7-day Follow-up Period After the First Vaccination (Administered at Day 1)
Description: Assessed solicited general adverse events are drowsiness, fever [defined as temperature equal to or above (>=) 38.degrees Celsius (C)/100.4 Fahrenheit (F) by any route], irritability/fussiness and loss of appetite. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, each of the active comparators and placebo groups separately as the study interest was to investigate solicited AEs during the follow-up period of RSV vaccine administration, compared to placebo and routine pediatric vaccines, especially comparing to the rates of Bexsero-related fever. As pre-specified in the protocol, the choice of active comparator or placebo was based on each participating country's standard of care.
Time Frame: During a 7-day follow-up period after the first vaccination (administered at Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Bexsero Group: Subjects received 3 doses of GSK's multicomponent meningococcal B vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
- Nimenrix Group: Subjects received 3 doses of Pfizer's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Days 1, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 31 and 121).
- Synflorix Group: Subjects received 3 doses of GSK's pneumococcal polysaccharide conjugate vaccine (administered at Days 31, 61 and at the end of RSV season 1) and 2 doses of Placebo (administered at Day 1 and Day 121).
- Menveo Group: Subjects received 2 doses of GSK's meningococcal group A, C, W-135 and Y conjugate vaccine (administered at Day 31 and at the end of RSV season 1) and 2 doses of Placebo (administered at Days 1 and 61)
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Placebo Group | Bexsero Group | Nimenrix Group | Synflorix Group | Menveo Group
Number analyzed (Participants) | 65 | 71 | 22 | 28 | 1 | 1 | 12
Participants
  Any Drowsiness | 12 | 19 | 7 | 11 | 0 | 1 | 2
  Any Fever | 9 | 24 | 5 | 11 | 0 | 0 | 2
  Any Irritability/Fussiness | 25 | 31 | 9 | 20 | 0 | 1 | 4
  Any Loss of appetite | 12 | 17 | 8 | 12 | 0 | 0 | 2

4. Primary Outcome: Number of Subjects With Any Solicited General AEs During a 7-day Follow-up Period After the Second Vaccination (Administered at Day 31)
Description: Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, each of the active comparators and placebo groups separately as the study interest was to investigate solicited AEs during the follow-up period of RSV vaccine administration, compared to placebo and routine pediatric vaccines, especially comparing to the rates of Bexsero-related fever. As pre-specified in the protocol, the choice of active comparator or placebo was based on each participating country's standard of care.
Time Frame: During a 7-day follow-up period after the second vaccination (administered at Day 31)
Population: Analysis was performed on the Exposed set, which included all subjects with at least 1 study vaccine administration documented and diary card completed after second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Placebo Group | Bexsero Group | Nimenrix Group | Synflorix Group | Menveo Group
Number analyzed (Participants) | 63 | 71 | 20 | 27 | 1 | 1 | 12
Participants
  Any Drowsiness | 10 | 18 | 3 | 5 | 0 | 0 | 4
  Any Fever | 6 | 28 | 0 | 1 | 0 | 0 | 3
  Any Irritability/Fussiness | 18 | 33 | 3 | 9 | 0 | 0 | 6
  Any Loss of appetite | 7 | 22 | 3 | 4 | 0 | 0 | 4

5. Primary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AEs are reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: During a 30-day follow-up period across the 2 vaccinations administered at Day 1 and Day 31
Population: The analysis was performed on the Exposed set, which included all subjects with at least one study vaccine administration documented. Study interest was to check unsolicited AEs only during the follow-up period of study RSV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 34 | 45 | 36

6. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) From Day 1 up to Day 61
Description: Assessed serious adverse events (SAEs) include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Any = occurrence of SAE regardless of intensity grade or relation to study vaccination. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of theindividual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: From Day 1 up to Day 61
Population: The analysis was performed on the Exposed set, which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 3 | 3 | 0

7. Primary Outcome: Number of Subjects With Episode of Spontaneous or Excessive Bleeding (AE of Special Interest)
Description: Any episode of spontaneous or excessive bleeding if occurring after vaccination was to be fully investigated with a full range of hematological tests to identify the underlying cause and reported as an AE of special interest. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: During a 30-day follow-up period across the 2 vaccinations administered at Day 1 and Day 31
Population: The analysis was performed on the Exposed set, which included all subjects with at least one study vaccine administration documented. Study interest was to check episode of spontaneous or excessive bleeding (AE of special interest) only during the follow-up period of study RSV vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 1 | 0 | 0

8. Secondary Outcome: Number of Subjects With Respiratory Tract Infection Associated With RSV Infection (RSV-RTI), Lower Respiratory Tract Infection Associated With RSV Infection (RSV-LRTI), Severe RSV-LRTI and Very Severe RSV-LRTI (According to Standardized Case Definitions)
Description: According to standardized case definitions,RSV-RTI is a subject having runny nose/blocked nose/ cough & confirmed RSV infection.RSV-LRTI is a subject having history of cough/ difficulty breathing[based on history reported by parents] & blood oxygen saturation (SpO2) lower than(<)95 percent (%)/ respiratory rate (RR) increase & confirmed RSV infection Severe RSV-LRTI-Cases meeting RSV-LRTI case definition & an SpO2<93 %/lower chest wall in-drawing. Very severe RSV-LRTI-Cases meeting RSV-LRTI case definition & an SpO2<90%/inability to feed/failure to respond/unconscious.Analysis of this outcome measure was reported for RSV1D pooled, RSV2D pooled & comparator_placebo pooled groups as data was collected based on different standard of care provided at participating countries rather than randomization to each of the groups.Per the pre-specified analysis plan,data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups
Time Frame: From first vaccination (Day 1) up to the end of the first RSV transmission season (up to 1 year)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants
  RSV-RTI | 21 | 17 | 27
  RSV-LRTI | 3 | 3 | 4
  Severe RSV-LRTI | 1 | 1 | 3
  Very severe RSV-LRTI | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects With RSV-RTI, RSV-LRTI, Severe RSV-LRTI and Very Severe RSV-LRTI (According to Standardized Case Definitions)
Description: Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: From first vaccination (Day 1) up to the end of the second RSV transmission season (up to 2 years)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants
  RSV-RTI | 23 | 18 | 30
  RSV-LRTI | 3 | 3 | 4
  Severe RSV-LRTI | 1 | 1 | 3
  Very severe RSV-LRTI | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With SAEs From First Vaccination (Day 1) up to the End of the Second RSV Transmission Season (up to 2 Years)
Description: Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the 15 groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: From first vaccination (Day 1) up to the end of the second RSV transmission season (up to 2 years)
Population: The analysis was performed on the Exposed set, which includes all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 7 | 11 | 3

11. Secondary Outcome: Number of Subjects With RSV-LRTI (AE of Special Interest) From First Vaccination (Day 1) up to the End of the First RSV Transmission Season (up to 1 Year)
Description: Subjects experiencing an LRTI associated with RSV infection were reported as AE of special interest. To identify RSV-LRTI for the purpose of AE of specific interest, the diagnosis was based on the investigators' clinical judgment taking into account the clinical history, the examination, relevant medical investigations and locally-available diagnostic test for RSV. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: From first vaccination (Day 1) up to the end of the first RSV transmission season (up to 1 year)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 7 | 6 | 7

12. Secondary Outcome: Number of Subjects With RSV-LRTI (AE of Special Interest) From First Vaccination (Day 1) up to the End of the Second RSV Transmission Season (up to 2 Years)
Description: as for outcome 9
Time Frame: From first vaccination (Day 1) up to the end of the second RSV transmission season (up to 2 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 65 | 71 | 65
Participants | 7 | 6 | 7

13. Secondary Outcome: Number of RSV Infected Subjects With a Negative RSV Exposure Status (at Screening Based on In-stream Baseline Serological Testing) With Very Severe RSV-LRTI (According to Standardized Case Definition)
Description: Very severe RSV LRTI are cases meeting the case definition of RSV-LRTI AND a SpO2 <90%, OR inability to feed, OR failure to respond/unconscious. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: From first vaccination (Day 1) up to the end of the first RSV transmission season (up to 1 year)
Population: The analysis was performed on the Exposed set with a negative RSV exposure status, which included all vaccinated subjects assessed as RSV unexposed at screening based on in-stream baseline serological testing.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 49 | 58 | 52
Participants | 0 | 0 | 0

14. Secondary Outcome: Anti-RSV-A Neutralizing Antibody Titers
Description: Humoral response to the investigational RSV vaccine was measured in terms of anti-RSV-A neutralizing antibody titers and expressed as geometric mean titers (GMTs) in Estimated Dilution 60 (ED60) titers. Analysis of this outcome measure were reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: At pre-vaccination (Screening), Day 31, Day 61 and at the end of the first RSV transmission season (EOS1) (up to 1 year)
Population: The analysis was performed on the Per-protocol set for analysis of immunogenicity, which included all subjects with at least one study vaccine administration documented, who complied with eligibility criteria, study procedures up to the end of the study and had immunogenicity results for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 64 | 71 | 61
Titers
  Screening | 26.8 [20.7 to 34.6] | 29.6 [23.6 to 37.3] | 32.2 [24.9 to 41.6]
  Day 31: number analyzed (Participants) | 63 | 69 | 61
  Day 31 | 60.2 [44.2 to 81.9] | 116.2 [87.6 to 153.9] | 18.9 [14.8 to 24.1]
  Day 61: number analyzed (Participants) | 63 | 70 | 56
  Day 61 | 54.3 [37.7 to 78] | 259.4 [211.6 to 318.1] | 14.4 [11.8 to 17.7]
  EOS1: number analyzed (Participants) | 60 | 70 | 61
  EOS1 | 165 [95 to 286.6] | 223.7 [154.7 to 323.4] | 66.3 [40.2 to 109.5]

15. Secondary Outcome: Anti-RSV-F Antibody Concentrations
Description: Humoral response to the investigational RSV vaccine was measured in terms of anti-RSV-F antibody concentrations and expressed as geometric mean concentrations (GMCs) in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EU/mL). Analysis of this outcome measure was reported for the RSV1D pooled, RSV2D pooled, and comparator_placebo pooled groups as data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
Number analyzed (Participants) | 64 | 71 | 61
EU/mL
  Screening: number analyzed (Participants) | 63 | 71 | 61
  Screening | 93.1 [72.7 to 119.1] | 81.9 [61.8 to 108.6] | 86 [65.5 to 112.7]
  Day 31: number analyzed (Participants) | 64 | 70 | 60
  Day 31 | 2035.2 [1490 to 2779.9] | 4550.8 [3354.6 to 6173.7] | 46.2 [31.6 to 67.6]
  Day 61: number analyzed (Participants) | 61 | 70 | 55
  Day 61 | 1976.5 [1346.2 to 2901.8] | 9287.9 [7885.5 to 10939.7] | 24.6 [18.3 to 33]
  EOS1: number analyzed (Participants) | 60 | 69 | 60
  EOS1 | 5108.7 [3096.7 to 8428] | 4935.5 [3639.8 to 6692.4] | 345.1 [165.9 to 717.7]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period after any vaccination. Serious adverse events were collected from Day 1 up to the end of the second RSV transmission season (up to 2 years).
Description: Analysis of adverse events results were reported for the RSV 1D pooled, RSV 2D pooled, and comparator_placebo pooled groups as adverse events data collection was based on different standard of care provided at participating countries rather than randomization to each of the individual groups. According to the pre-specified analysis plan, data collected for participant flow, baseline characteristics and adverse events reporting were not analyzed for the individual groups.
Arm/Group | RSV1D Pooled Group | RSV2D Pooled Group | Comparator_Placebo Pooled Group
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/71 | 0/65
Serious Adverse Events (participants affected / at risk) | 7/65 | 11/71 | 3/65
Other Adverse Events (participants affected / at risk) | 57/65 | 67/71 | 57/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV1D Pooled Group (N=65) | RSV2D Pooled Group (N=71) | Comparator_Placebo Pooled Group (N=65)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV1D Pooled Group (N=65) | RSV2D Pooled Group (N=71) | Comparator_Placebo Pooled Group (N=65)
Pyrexia (General disorders) | 17 (18) | 37 (54) | 23 (25)
Administration site erythema (General disorders) | 9 (13) | 11 (13) | 26 (33)
Administration site pain (General disorders) | 13 (16) | 12 (19) | 19 (24)
Administration site swelling (General disorders) | 3 (3) | 4 (6) | 18 (19)
Injection site bruising (General disorders) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (14) | 13 (15) | 15 (19)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 8 (11) | 5 (5)
Gastroenteritis (Infections and infestations) | 3 (3) | 7 (7) | 2 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 34 (44) | 41 (65) | 36 (53)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 17 (19) | 32 (39) | 25 (33)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 18 (22) | 29 (37) | 26 (33)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (5) | 2 (2)
Teething (Gastrointestinal disorders) | 4 (4) | 4 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital pulmonary valve atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03636906/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03636906/SAP_001.pdf